CLINICAL TRIAL: NCT03289221
Title: Effects of High-Intensity Focused Ultrasound (HIFU) Treatment on Fecal Continence and Anorretal Fisiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Transplante Doutor Euryclides de Jesus Zerbini (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HIFU02
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Anal Continence After High-Intensity Focused Ultrasound (HIFU) Treatment

STUDY DESIGN:
Intervention Model Description: Thirty (30) consecutive patients indicated for treatment of prostate cancer with HIFU (FocalOneR, Edap TMS, France) will be selected to the manometry study before the treatment together with the application of specific questionnaires (Cleveland Clinic Incontinence Score-CCIS, Fecal Incontinence Quality of Life Score-FIQLS, and Rome IV for functional constipation. This evaluaton will be conducted again after the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Thirty (30) consecutive patients indicated for treatment of prostate cancer with HIFU (FocalOneR, Edap TMS, France) will be selected to the manometry study before the treatment together with the application of specific questionnaires (Cleveland Clinic Incontinence Score-CCIS, Fecal Incontinence Quality of Life Score-FIQLS, and Rome IV for functional constipation. This evaluaton will be conducted again after the treatment.
  Interventions: Diagnostic Test: Anal Manometry

INTERVENTIONS:
Diagnostic Test: Anal Manometry — A suppository will be used to clean the rectum 3 to 4 hours prior to the examination. And the pressures of rest and voluntary contraction of the anal sphincter will be evaluated, as well as the behavior of the pubortal muscle during the evacuation maneuver. Retinal inhibitory reflex (RIRA), sensitivity and rectal capacity will also be evaluated.
  Questionnaires that evaluate the pre and post HIFU anal physiology will also be applied at the time of manometry.

SUMMARY:
Investigate the presence of hypotonic anal sphincter after anorectal dilatation and High-Intensity Focused Ultrasound (HiFU) , through the aplication of questionnaires and Anorectal Manometry before and after this treatment.

DETAILED DESCRIPTION:
Primary Investigate the presence of hypotonic anal sphincter after anorectal dilatation and HiFU procedure

Secondary

1. Detect the presence of fecal incontinence
2. Demonstrate the absence of alterations in the fecal pattern
3. Detect alterations in rectal filling sensation and e evacuation desire
4. Evaluate anal pain

PATIENTS AND METHODS Thirty (30) consecutive patients indicated for treatment of prostate cancer with HIFU (FocalOneR, Edap TMS, France) will be selected. The specific inclusion and exclusion criteria are specified below. All should present the diagnosis of usual acinar adenocarcinoma of prostate Gleason score 6 (3 + 3) or Gleason 7 (3 + 4). No patient may have PSA greater than 10.0. A digital prostate exam should show prostate-restricted disease. The clinical staging should be ≤ cT2a. There will be no age limit for inclusion. Patients may not have anatomical, functional or pathological alterations of the anal canal and rectus or history of anorectal trauma and may not have a diagnosis of psychoneurologic diseases, such as: Depression, Stroke, Schizophrenia, Degenerative Neurological Diseases or others.

All patients will be submitted to the manometry study the week prior to HIFU together with the application of specific questionnaires (Cleveland Clinic Incontinence Score-CCIS, Fecal Incontinence Quality of Life Score-FIQLS, and Rome IV for functional constipation. This examination will be conducted in a friendly environment and by experienced professionals.

Patients who met the inclusion and exclusion criteria and who signed the informed consent form will be linked to the study.

REALIZATION OF HIFU, MANOMETRY AND QUESTIONNAIRES All patients treated with HIFU should have prostate volume less than 40g for treatment of hemigland or 30g for whole gland treatments. Patients will have rectal cleansing for 3 to 6 hours prior to the procedure and will be treated according to the FocalOneR treatment protocol, with general anesthesia and bladder catheterization with Foley 16 or 18 Fr catheter. After general anesthesia and positioning, digital dilatation of the anal sphincter and introduction of the HIFU probe will be performed. With the end of treatment, the probe is withdrawn, and the patient awake from the anesthesia. In the anesthetic recovery room will be applied the visual pain scale that will also be applied at the time of hospital discharge and on the thirtieth day of the procedure. Patients may receive common analgesics as needed.

To perform the manometry examination it is necessary that the patient is awake, without effect of sedatives and cooperating with examination. A suppository will be used to clean the rectum 3 to 4 hours prior to the examination. And the pressures of rest and voluntary contraction of the anal sphincter will be evaluated, as well as the behavior of the pubortal muscle during the evacuation maneuver. Retinal inhibitory reflex (RIRA), sensitivity and rectal capacity will also be evaluated.

Questionnaires that evaluate the pre and post HIFU anal physiology will also be applied at the time of manometry.

PLACE OF ACHIEVEMENT OF RESEARCH AND FINANCIAL RESOURCES The selected patients will perform the tests of manometry, the HIFU procedure, the follow-up and treatment of possible complications in the Hospital of Transplants Euryclides de Jesus Zerbini (Hospital Brigadeiro) through the Unique Health System (UHS/SUS). This research does not have any private financial support. The funds will come from the SUS and there will be no excess expenses to the SUS.

THE SAMPLE AND TIME OF RECRUITMENT Thirty (30) consecutive patients will be selected, with indication of treatment of malignant neoplasm of the prostate by the HIFU method, and that they respect the criteria of inclusion and exclusion. The estimated time for recruitment of the completed sample is 30 days. And the deadline for the entire study will be 60 days from the start of the study.

STATISTIC Statistical analysis will be performed with the help of SPSS 17.0 for Windows. Results such as mean, median and prevalence will be calculated. The significance level adopted will be 0.05.

COSTS All manometry examinations will be performed at the Paulista Endoscopy Center (CPE - CNPJ: 48.109.011 / 0001-30). The CPE will make available all the physical structure, employees, trained doctors and materials needed to perform the manometry exams. Patients will be asked to attend CPE (Rua Cincinato Braga, 37, CJ. 12, 1st floor, Bela Vista, SP) and NO COST TO THE BRIGADEIRO HOSPITAL, FOR PATIENTS AND / OR RESEARCHERS.

RISK ANALYSIS, PROTECTION MEASURES AND SUSPENSION OF RESEARCH This research does not involve any experimental procedure. The treatment of patients with HIFU is already established with specific cancer survival results found in the literature for 10 years (7, 8).

The manometry exam is a very safe technique and practically free of complications. In very rare cases, small rectal bleeding of spontaneous resolution, low intensity pain in the anal region, and very rarely, perforation of the rectal mucosa may occur with the need for surgery. (19) In any case, the presence of complications will be treated at the Brigadeiro Hospital, which has urologists 24 hours a day, 7 days a week. In addition, the Brigadeiro Hospital has emergency room for patients 24/7 with clinicians on call and support general surgery staff. The patients will be instructed to return immediately to the Hospital in case of any complications, where they will be attended by a doctor of the urology team and communicated the occurrence to the researchers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of any age with diagnosis of usual acinar adenocarcinoma of the prostate;
2. Patients that treatment with HIFU is an option;
3. And, that they accept to undergo the pre-and post-HIFU anorectal manometry;
4. And, answer the questionnaires applied;
5. And, signature of the informed consent form.

Exclusion Criteria:

1. Patients who have no indication of HIFU treatment;
2. Or, who have already undergone some anorectal surgery;
3. Or, that they present some psychoneurological disease;
4. Or, who have anatomical, functional or pathological alterations of the rectum or anal;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Anal sphicter evaluation | 2 months
  Investigate the presence of hypotonic anal sphincter after anorectal dilatation and HiFU procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jose RC Silvino, Principal Investigator — Euryclides de Jesus Zerbini Transplant Hospital
Locations (1):
- Euryclides de Jesus Zerbini Transplant Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Crawford ED. Epidemiology of prostate cancer. Urology. 2003 Dec 22;62(6 Suppl 1):3-12. doi: 10.1016/j.urology.2003.10.013. PMID 14706503
- [Result] Carter HB, Pearson JD. Prostate-specific antigen testing for early diagnosis of prostate cancer: formulation of guidelines. Urology. 1999 Nov;54(5):780-6. doi: 10.1016/s0090-4295(99)00271-x. No abstract available. PMID 10565733
- [Result] Jemal A, Ward EM, Johnson CJ, Cronin KA, Ma J, Ryerson B, Mariotto A, Lake AJ, Wilson R, Sherman RL, Anderson RN, Henley SJ, Kohler BA, Penberthy L, Feuer EJ, Weir HK. Annual Report to the Nation on the Status of Cancer, 1975-2014, Featuring Survival. J Natl Cancer Inst. 2017 Sep 1;109(9):djx030. doi: 10.1093/jnci/djx030. PMID 28376154
- [Result] D'Amico AV, Whittington R, Malkowicz SB, Schultz D, Blank K, Broderick GA, Tomaszewski JE, Renshaw AA, Kaplan I, Beard CJ, Wein A. Biochemical outcome after radical prostatectomy, external beam radiation therapy, or interstitial radiation therapy for clinically localized prostate cancer. JAMA. 1998 Sep 16;280(11):969-74. doi: 10.1001/jama.280.11.969. PMID 9749478
- [Result] Gelet A, Chapelon JY, Bouvier R, Souchon R, Pangaud C, Abdelrahim AF, Cathignol D, Dubernard JM. Treatment of prostate cancer with transrectal focused ultrasound: early clinical experience. Eur Urol. 1996;29(2):174-83. PMID 8647143
- [Result] Thuroff S, Chaussy C. Evolution and outcomes of 3 MHz high intensity focused ultrasound therapy for localized prostate cancer during 15 years. J Urol. 2013 Aug;190(2):702-10. doi: 10.1016/j.juro.2013.02.010. Epub 2013 Feb 13. PMID 23415962
- [Result] Crouzet S, Chapelon JY, Rouviere O, Mege-Lechevallier F, Colombel M, Tonoli-Catez H, Martin X, Gelet A. Whole-gland ablation of localized prostate cancer with high-intensity focused ultrasound: oncologic outcomes and morbidity in 1002 patients. Eur Urol. 2014 May;65(5):907-14. doi: 10.1016/j.eururo.2013.04.039. Epub 2013 Apr 30. PMID 23669165
- [Result] Ramsay CR, Adewuyi TE, Gray J, Hislop J, Shirley MD, Jayakody S, MacLennan G, Fraser C, MacLennan S, Brazzelli M, N'Dow J, Pickard R, Robertson C, Rothnie K, Rushton SP, Vale L, Lam TB. Ablative therapy for people with localised prostate cancer: a systematic review and economic evaluation. Health Technol Assess. 2015 Jul;19(49):1-490. doi: 10.3310/hta19490. PMID 26140518
- [Result] van Velthoven R, Aoun F, Marcelis Q, Albisinni S, Zanaty M, Lemort M, Peltier A, Limani K. A prospective clinical trial of HIFU hemiablation for clinically localized prostate cancer. Prostate Cancer Prostatic Dis. 2016 Mar;19(1):79-83. doi: 10.1038/pcan.2015.55. Epub 2015 Nov 24. PMID 26597660
- [Result] Feijoo ER, Sivaraman A, Barret E, Sanchez-Salas R, Galiano M, Rozet F, Prapotnich D, Cathala N, Mombet A, Cathelineau X. Focal High-intensity Focused Ultrasound Targeted Hemiablation for Unilateral Prostate Cancer: A Prospective Evaluation of Oncologic and Functional Outcomes. Eur Urol. 2016 Feb;69(2):214-20. doi: 10.1016/j.eururo.2015.06.018. Epub 2015 Jul 9. PMID 26164416
- [Result] Peltier A, Aoun F, Lemort M, Kwizera F, Paesmans M, Van Velthoven R. MRI-targeted biopsies versus systematic transrectal ultrasound guided biopsies for the diagnosis of localized prostate cancer in biopsy naive men. Biomed Res Int. 2015;2015:571708. doi: 10.1155/2015/571708. Epub 2015 Jan 27. PMID 25692142
- [Result] Perry RE, Blatchford GJ, Christensen MA, Thorson AG, Attwood SE. Manometric diagnosis of anal sphincter injuries. Am J Surg. 1990 Jan;159(1):112-6; discussion 116-7. doi: 10.1016/s0002-9610(05)80615-4. PMID 2294787
- [Result] Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97. doi: 10.1007/BF02050307. PMID 8416784
- [Result] Rockwood TH, Church JM, Fleshman JW, Kane RL, Mavrantonis C, Thorson AG, Wexner SD, Bliss D, Lowry AC. Fecal Incontinence Quality of Life Scale: quality of life instrument for patients with fecal incontinence. Dis Colon Rectum. 2000 Jan;43(1):9-16; discussion 16-7. doi: 10.1007/BF02237236. PMID 10813117
- [Result] Williams N, Barlow J, Hobson A, Scott N, Irving M. Manometric asymmetry in the anal canal in controls and patients with fecal incontinence. Dis Colon Rectum. 1995 Dec;38(12):1275-80. doi: 10.1007/BF02049152. PMID 7497839
- [Result] Taylor BM, Beart RW Jr, Phillips SF. Longitudinal and radial variations of pressure in the human anal sphincter. Gastroenterology. 1984 Apr;86(4):693-7. PMID 6698369
- [Result] Nelson R, Norton N, Cautley E, Furner S. Community-based prevalence of anal incontinence. JAMA. 1995 Aug 16;274(7):559-61. PMID 7629985
- [Result] Jorge JM, Wexner SD. Anorectal manometry: techniques and clinical applications. South Med J. 1993 Aug;86(8):924-31. doi: 10.1097/00007611-199308000-00016. PMID 8351556